CLINICAL TRIAL: NCT06854900
Title: Investigation of Core Muscle Strength in Women with Primary Dysmenorrhoea
Brief Title: Core Muscle Strength in Women with Primary Dysmenorrhoea
Status: Completed | Type: Observational
Sponsor: Derya Azim (Other)
Responsible Party: Sponsor-Investigator, Derya Azim, Asst. Prof., Bandırma Onyedi Eylül University
Organization: Bandırma Onyedi Eylül University (Other)
Other Study IDs: 03. 04. 2024-176
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Pelvic Floor Muscle Weakness; Dysmenorrhea; Posture
Keywords: Pelvic floor; Dysmenorrhea; Posture; Core; Electromyography
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Dysmenorrhea: Dysmenorrhea
- Healthy Woman: Healthy Woman

SUMMARY:
The aim of this study is to compare core muscle strength, core muscle activations, and pelvic tilt angles in women with and without Primary Dysmenorrhea (PD).

DETAILED DESCRIPTION:
The study included 27 women with PD and 27 healthy women without primary dysmenorrhea. Demographic and menstrual information of the participants was recorded. The "Sport-Specific Core Muscle Strength & Stability Plank Test" protocol was applied to evaluate the core muscle strength of the participants. Pelvic floor, transversus abdominis, and multifidus muscle activations were assessed using the NeuroTrac® MyoPlus 2 dual-channel EMG ETS device. Pelvic tilt measurement was performed using the Apecs-AI Posture Assessment and Correction System®. Menstrual pain and symptoms were evaluated using the Menstrual Symptom Scale.

This study found that women with PD had higher muscle activations, lower pelvic tilt angles, and more severe menstrual symptoms. We believe these results may contribute to the etiology of PD.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria to be included in the study:

Age between 18 and 35 years

Diagnosed with Primary Dysmenorrhea (PD) according to the PD consensus criteria, which include:

Presence of menstrual pain within the first few years after menarche A Visual Analog Scale (VAS) pain score of 4 or higher in the last six months No pelvic pathology Having a regular menstrual cycle (21-35 days) No uterine disorders

Exclusion Criteria:

The sample size for the study was determined using the G*Power software (latest version 3.1.9.7; Heinrich-Heine-Universität Düsseldorf, Düsseldorf, Germany).

Since our study consists of two groups (participants with and without Primary Dysmenorrhea), the power analysis was conducted using the "Means: Difference between two independent means (two groups)" method.

Based on similar studies, an effect size of d = 0.726 was used for the calculation.

With a statistical power of 80% and a significance level of 5% (α = 0.05), the minimum required sample size was determined to be at least 25 participants per group, totaling 50 participants.Pregnancy or suspicion of pregnancy Active sexual life History of childbirth Use of an intrauterine device (IUD) History of surgery involving the abdomen, spine, or pelvic region within the last year Diagnosis of secondary dysmenorrhea Body mass index (BMI) of 30 or higher

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The sample size for the study was determined using the G*Power software (latest version 3.1.9.7; Heinrich-Heine-Universität Düsseldorf, Düsseldorf, Germany).
  Since our study consists of two groups (participants with and without Primary Dysmenorrhea), the power analysis was conducted using the "Means: Difference between two independent means (two groups)" method.
  Based on similar studies, an effect size of d = 0.726 was used for the calculation.
  With a statistical power of 80% and a significance level of 5% (α = 0.05), the minimum required sample size was determined to be at least 25 participants per group, totaling 50 participants.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 10 minutes
  One of the most commonly used methods for determining pain intensity is the Visual Analog Scale (VAS). In addition to assessing the severity of pain, VAS also provides information about how badly the patient feels due to pain. VAS consists of a 10 cm long line drawn either on a vertical or horizontal axis. At one end of the line, the phrase "no pain" is written, while at the other end, "unbearable pain" is indicated. Patients are asked to mark the point on the line that corresponds to the intensity of their pain. The distance from the "no pain" point to the patient's mark is then measured. This measurement provides a numerical value for the patient's pain intensity:
  0-2 cm: No pain 3-4 cm: Mild pain 5-6 cm: Moderate pain 7-8 cm: Severe pain 9-10 cm: Unbearable pain
Menstrual Symptom Scale | 15 minutes
  Developed by Chesney and Tasto (1975) to assess menstrual pain and symptoms, this scale was validated and tested for reliability by Güvenç et al. (2014). The scale consists of 22 items and is structured as a five-point Likert-type measure.
  Items 1-13 belong to the "Negative Effects/Somatic Complaints" subscale. Items 14-19 belong to the "Menstrual Pain Symptoms" subscale. Items 20-22 belong to the "Coping Methods" subscale. The Menstrual Symptom Scale score is calculated by taking the average total score of the items. Participants are asked to rate their menstrual symptoms by selecting a number between 1 (Never) and 5 (Always). A higher average score indicates greater severity of menstrual symptoms.
  Each subscale score is calculated by taking the average of the items within that subscale, and an increase in the subscale score reflects an increase in the severity of menstrual symptoms related to that specific subscale.
  The Cronbach's Alpha value of the scale is 0.86, indicating a hi
Core Strength Test | 20 minutes
  To assess participants' core muscle strength, the "Sport-Specific Core Muscle Strength & Stability Plank Test" protocol will be applied. This test was developed by Brian Mackenzie and its validity and reliability were studied by Tong et al. (2013) (95%, 0.94-0.99). The test consists of 8 steps and is performed against time, with a total duration of 3 minutes.
  Test Procedure:
  Step 1: The athlete assumes the plank position, and the test starts using a stopwatch. The athlete must hold this position for 60 seconds.
  Step 2: While maintaining the plank position, the athlete extends their right arm forward and holds it for 15 seconds.
  Step 3: The athlete extends their left arm forward and holds it for 15 seconds. Step 4: The athlete lifts their right foot 30 cm off the ground and holds it for 15 seconds.
  Step 5: The athlete lifts their left foot 30 cm off the ground and holds it for 15 seconds.
  Step 6: The athlete lifts their right arm and left foot simultaneously and holds them for 15 seco
Measurement of Core Muscle Strength Using Surface EMG | 30 minutes
  The strength of the pelvic floor, transversus abdominis, and multifidus muscles will be assessed using surface electromyography (sEMG). For this evaluation, the NeuroTrac® MyoPlus 2 dual-channel EMG ETS device (Verity Medical Ltd., UK) will be used to measure and record muscle activation. The device connects to a computer via specialized software.
  Electrode Placement and Preparation
  Electrodes:
  32 mm diameter, circular, adhesive silver-silver chloride (Ag-AgCl) electrodes will be used to measure muscle activity.
  Each participant will be provided with three personalized electrodes for the measurement.
  Skin Preparation:
  To ensure optimal signal quality, the skin area where the electrodes will be applied must be clean.
  Participants will be informed about preparing the application site before the measurement.
  To reduce skin impedance, the area where the surface electrodes will be placed will be cleaned with an alcohol wipe before the measurement.
  Electrode Placement for Pelvic Floor Musc

CONTACTS AND LOCATIONS:
Locations (1):
- Derya, Bandırma, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No